CLINICAL TRIAL: NCT02930304
Title: Non-Surgical Treatment Approaches in Patients With Newly Diagnosed Lateral Epicondylitis: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Eraslan, MSc, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO13/493
Record Dates: First submitted 2016-10-02; First posted 2016-10-12 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Tennis Elbow
Keywords: tennis elbow; pain; shock wave; kinesio taping
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Physical Therapy Modalities; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- first physiotherapy (Experimental): cold pack, TENS, exercise
  Interventions: Other: first physiotherapy
- second physiotherapy (Experimental): cold pack, TENS, exercise, kinesiotaping
  Interventions: Other: second physiotherapy
- third physiotherapy (Experimental): cold pack, TENS, ESWT, exercise
  Interventions: Other: third physiotherapy

INTERVENTIONS:
Other: first physiotherapy — physiotherapy program consists of cold pack, Transcutaneous electrical nerve stimulation (TENS), and home exercise programme including stretching and eccentric strength exercises will be applied five times a week total 15 sessions
  Other Names: physiotherapy
  Arms: first physiotherapy
Other: second physiotherapy — physiotherapy program consists of cold pack, Transcutaneous electrical nerve stimulation (TENS), and home exercise programme including stretching and eccentric strength exercises will be applied five times a week total 15 sessions. Kinesio taping will be applied two times per week total six times in addition to conventional physiotherapy
  Other Names: kinesiotaping
  Arms: second physiotherapy
Other: third physiotherapy — physiotherapy program consists of cold pack, Transcutaneous electrical nerve stimulation (TENS), and home exercise programme including stretching and eccentric strength exercises will be applied five times a week total 15 sessions. Extracorporeal shockwave therapy (ESWT) will be applied one times per week total three session.
  Other Names: Extracorporeal shockwave therapy (ESWT)
  Arms: third physiotherapy

SUMMARY:
Lateral epicondylitis (tennis elbow) is a painful musculoskeletal condition, which is considered to be due to overuse, over-stress or over-exertion of the wrist extensors of the forearm, especially extensor carpi radialis brevi.

The aim of this study is to The compare the short-term effects of different physiotherapy approaches on pain, function and grip strength in the rehabilitation of patients with lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis (tennis elbow) is a painful musculoskeletal condition, which is considered to be due to overuse, over-stress or over-exertion of the wrist extensors of the forearm, especially extensor carpi radialis brevi. Different treatment approaches are described in the literature. The primary aim of the treatment approaches are decrease the pain and improve the functional level in patients with lateral epicondylitis. Thus, decreasing pain and regaining the functional performance in the daily living activity is essential in early diagnosed patients.

The aim of this study is to compare the short-term effects of different treatment approaches on pain, function and grip strength in the rehabilitation of patients with lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with tennis elbow,
* and the duration of symptoms was between 8 and 10 weeks,
* and pain over the lateral epicondyle, pain during grip strength testing, and pain with one of the following tests: extensor carpi radialis test (i.e., resisted middle-finger extension), resisted wrist extension, or passive stretch of the wrist extensors.
* Furthermore, the participants had to agree to abstain from any other form of treatment during their involvement in this study

Exclusion Criteria:

* patients with inflammatory, autoimmune, endocrine or kidney diseases, cubital tunnel syndrome, carpal tunnel syndrome, radiculopathies due to cervical disc pathologies, additional shoulder-hand-wrist pathologies, inflammatory arthritis, upper extremity operations or traumas,
* allergies to adhesive tape,
* and the patients who received corticosteroid injection due to lateral epicondylitis within the last 3 months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
pain assessment | from baseline to third week after treatment sessions
  pain intensity will de assessed by using Visual Analog Scale at rest, activity and at night. All assessment will be recorded at baseline and at the end of the three week treatment sessions

SECONDARY OUTCOMES:
functional assessment | from baseline to third week after treatment sessions
  functional status will be assessed by using Patient-Rated Tennis Elbow Evaluation Scale (PRTEE). All assessment will be recorded at baseline and at the end of the three week treatment sessions
maximum grip strength evaluation | from baseline to third week after treatment sessions
  maximum grip strength will be assessed with hand dynamometer both elbow flexion and extension position. All assessment will be recorded at baseline and at the end of the three week treatment sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Dept. of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No